CLINICAL TRIAL: NCT04833894
Title: Open-label Uncontrolled Trial to Evaluate Pharmacokinetics, Pharmacodynamics, Safety, and Activity of Efgartigimod in Children From 2 to Less Than 18 Years of Age With Generalized Myasthenia Gravis
Brief Title: Evaluating the Pharmacokinetics, Pharmacodynamics, and Safety of Efgartigimod Administered Intravenously in Children With Generalized Myasthenia Gravis
Acronym: ADAPT Jr
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-2006; 2024-513854-31-00 (EU CTIS Number)
Record Dates: First submitted 2021-03-16; First posted 2021-04-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Efgartigimod (Experimental): Patients receiving efgartigimod intravenous (IV) treatment
  Interventions: Biological: Efgartigimod IV

INTERVENTIONS:
Biological: Efgartigimod IV — Intravenous infusion of Efgartigimod

SUMMARY:
The purpose of this trial is to investigate the PK, PD, safety, and activity of efgartigimod IV in children and adolescents aged from 2 to less than 18 years of age with gMG.

Trial details include:

* The maximum trial duration for each individual participant will be approximately 28 weeks
* The treatment duration will be 8 weeks for the dose-confirmatory part (Part A) and 18 weeks for the treatment response-confirmatory part (Part B)

ELIGIBILITY:
Inclusion Criteria:

1. Ability of the participant and/or his/her legally authorized representative to understand the requirements of the trial and provide written informed consent/assent, if applicable (including consent/assent for the use and disclosure of research-related health information), willingness and ability to comply with the trial protocol procedures (including attending the required trial visits).
2. Male or female participants between 2 to less than 18 years of age at the time of providing informed consent/assent. Age groups are enrolled in a staggered fashion respectively: 6 participants in the 12 to less than 18 years of age group followed by 6 participants in the 2 to less than 12 years of age group at the time of providing informed consent/assent.
3. Diagnosed with Generalized Myasthenia Gravis (gMG) with confirmed documentation
4. Meeting the clinical criteria as defined by the Myasthenia Gravis Foundation of America (MGFA) class II, III, and IVa.
5. Eligible participants should have an unsatisfactory response (efficacy and/or safety) to immunosuppressants, steroids or acetylcholinesterase (AChE) inhibitors and should be on stable concomitant gMG therapy of adequate duration before screening.
6. Positive serologic test for acetylcholine receptor (anti-AChR) antibodies at screening (for younger participants (<15kg) historical values can be used).
7. Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical trials. A subject is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active.

   1. Male participants: Male participants must agree to not donate sperm from of providing informed consent/assent until they have completed the trial.
   2. Female participants: Female adolescents of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline before investigational medicinal product (IMP) can be administered.

Exclusion Criteria:

1. Participants with MGFA class I, IVb, and V.
2. Female adolescents of childbearing potential: Pregnancy or lactation, or the participant intends to become pregnant during the trial or within 90 days after the last dose of IMP.
3. Has any of the following medical conditions:

   1. Clinically significant uncontrolled active or chronic bacterial, viral, or fungal infection at screening.
   2. Any other known autoimmune disease that, in the opinion of the investigator, would interfere with an accurate assessment of clinical symptoms of myasthenia gravis or put the participant at undue risk.
   3. History of malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥3 years before the first administration of IMP. Participants with the following cancers can be included at any time: Adequately treated basal cell or squamous cell skin cancer; Carcinoma in situ of the cervix; Carcinoma in situ of the breast; Incidental histological findings of prostate cancer
   4. Clinical evidence of other significant serious diseases, or have had a recent major surgery, or who have any other condition that, in the opinion of the investigator, could confound the results of the trial or put the participant at undue risk
4. Worsening muscle weakness secondary to concurrent infections or medications (aminoglycosides, fluoro-quinolones, beta-blockers, etc).
5. A documented lack of clinical response to plasma exchange (PLEX).
6. Received a live or live-attenuated vaccine fewer than 28 days before screening. Receiving an inactivated, subunit, polysaccharide, or conjugate vaccine any time before screening is not exclusionary.
7. Received a thymectomy <3 months before screening or 1 is planned to be performed during the trial period.
8. The following results from these diagnostic assessments will be considered exclusionary:

   a. Positive serum test at screening for an active viral infection with any of the following conditions: Hepatitis B virus (HBV) that is indicative of an acute or chronic infection; Hepatitis C virus (HCV) based on HCV antibody assay; Positive HIV serology at screening; Positive nasopharyngeal swab polymerase chain reaction (PCR) test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at screening.
9. Using the following prior or concomitant therapies: Use of an investigational product within 3 months or 5 half-lives (whichever is longer) before the first dose of IMP, Use of any monoclonal antibody within the 6 months before the first dose of IMP, Use of intravenous immunoglobulin (IVIg), administered subcutaneously or intramuscularly, or PLEX within 4 weeks before screening.
10. Total immunoglobulin (IgG) levels <6 g/L below the lower limit of normal (LLN) according to the reference ranges of the central laboratory for participant by sex and age at screening.
11. A known hypersensitivity reaction to efgartigimod or any of its excipients.
12. Current participation in another interventional clinical trial or previous participation in an efgartigimod trial with at least 1 dose of IMP received.
13. History (within 12 months of screening) of current alcohol, drug, or medication abuse as assessed by the investigator.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Efgartigimod concentrations as input for compartmental, model-driven analysis to determine (age and size dependency of) Clearance (CL) | up to 26 weeks
  Blood samples will be collected from each participant for measurement of serum concentrations of efgartigimod
Efgartigimod concentrations as input for compartmental, model-driven analysis to determine (age and size dependency of) Volume of Distribution (Vd) | up to 26 weeks
  Blood samples will be collected from each participant for measurement of serum concentrations of efgartigimod
Total Immunoglobulin G (IgG) levels as input for pharmacokinetics (PK) and pharmacodynamics (PD) modeling analysis | up to 26 weeks
  Total Immunoglobulin G levels will be measured from blood samples
Anti-acetylcholine receptors antibodies (AChR-Ab) as input for pharmacokinetics (PK) and pharmacodynamics (PD) modeling analysis | up to 26 weeks
  Total Immunoglobulin G (IgG) levels will be measured from blood samples

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESIs) | up to 28 weeks
Efgartigimod serum concentrations from blood samples | up to 26 weeks
Absolute values of levels of total Immunoglobulin G (IgG) from blood samples | up to 26 weeks
Change from baseline of levels of total Immunoglobulin G (IgG) from blood samples | up to 26 weeks
Percentage change from baseline of total Immunoglobulin G (IgG) from blood samples | up to 26 weeks
Absolute values of anti-acetylcholine receptor antibodies (AChR-Ab) from blood samples | up to 26 weeks
Change from baseline of anti-acetylcholine receptor antibodies (AChR-Ab) from blood samples | up to 26 weeks
Percentage change from baseline of anti-acetylcholine receptor antibodies (AChR-Ab) from blood samples | up to 26 weeks
Incidence of anti-drug antibodies (ADAs) against efgartigimod in serum samples | up to 28 weeks
Prevalence of anti-drug antibodies (ADAs) against efgartigimod in serum samples | up to 28 weeks
Absolute values of total Myasthenia Gravis Activity of Daily Living (MG-ADL) score. Total score can range from 0 to 24, with higher total scores indicating more impairment. | up to 26 weeks
Change from baseline of total Myasthenia Gravis Activity of Daily Living (MG-ADL) score. Total score can range from 0 to 24, with higher total scores indicating more impairment. | up to 26 weeks
Absolute values of total Quantitative Myasthenia Gravis Score (QMG score). The total possible score is 39, where higher total scores indicate more severe impairments. | up to 26 weeks
Change from baseline of total Myasthenia Gravis Score (QMG score). The total possible score is 39, where higher total scores indicate more severe impairments. | up to 26 weeks
Absolute values of total score EuroQoL 5 Dimensions Youth (EQ-5D-Y) | up to 26 weeks
  Description of the participant's health state is done by digits for 5 dimensions combined in a 5-digit number. A unique health state is defined by combining 1 level from each of the 5 dimensions. Each state is referred to in terms of a 5-digit code, whereas code 11111 would indicate no problems in any of the 5 dimensions and 33333 would indicate worst problems in any of the 5 dimensions.
Change from baseline of total score EuroQoL 5 Dimensions Youth (EQ-5D-Y) | up to 26 weeks
  Description of the participant's health state is done by digits for 5 dimensions combined in a 5-digit number. A unique health state is defined by combining 1 level from each of the 5 dimensions. Each state is referred to in terms of a 5-digit code, whereas code 11111 would indicate no problems and 33333 would indicate worst problems in any of the 5 dimensions.
Values of Neurological Quality of Life (Neuro-QoL) pediatric fatigue questionnaire | up to 26 weeks
Change from baseline of Neurological Quality of Life (Neuro-QoL) pediatric fatigue questionnaire | up to 26 weeks
Change in protective antibody titers to vaccines received before or during the trial from blood samples | up to 28 weeks

CONTACTS AND LOCATIONS:
Locations (24):
- United States (3):
  - Ann and Robert H Lurie Children's Hospital of Chicago - Main Hospital, Chicago, Illinois
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Virginia (UVA) Health - Developmental Pediatrics Clinic, Charlottesville, Virginia
- Medizinische Universitat Wien, Vienna, Austria
- Universitair Ziekenhuis Antwerpen, Antwerp, Belgium
- British Columbia Children's Hospital, Vancouver, Canada
- France (2):
  - AP-HM - Hopital de la Timone, Marseille
  - Assistance Publique Hopitaux de Paris (AP-HP) - Hopital Necker-Enfants Malades, Paris
- Georgia (2):
  - Vian - M. Iashvili Children's Central Hospital, Tbilisi
  - Tbilisi State Medical University - Givi Zhvania Pediatric Academic Clinic, Tbilisi
- Germany (2):
  - Charite Universitaetsmedizin Berlin - Campus Virchow-Klinikum - Sozialpadiatrisches Zentrum, Berlin
  - Universitätsklinikum Essen, Essen
- Italy (3):
  - Azienda Ospedaliera Universitaria Policlinico Consorziale Di Bari, Bari
  - Azienda Ospedaliero Universitaria A. Meyer, Florence
  - Ospedale Giannina Gaslini, Genova
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Woj. Pomorskie
  - Wielospecjalistyczna Poradnia Lekarska Synapsis, Katowice, Woj. Slaskie
  - Centralny Szpital Kliniczny - Uniwersyteckie Centrum Kliniczne WUM, Warsaw
- Spain (2):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- United Kingdom (3):
  - Great Ormand Street Hospital for Children NHS Foundation Trust - Great Ormond Street Hospital, London
  - Manchester University NHS Foundation Trust - Royal Manchester Children's Hospital, Manchester
  - Oxford University Hospitals NHS Foundation Trust - John Radcliffe Hospital Children's Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Undecided